CLINICAL TRIAL: NCT02676544
Title: Prostate Embolization for Massive Benign Prostatic Hypertrophy (BPH)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Device approved for this use
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Albert Scappaticci, PhD, MD, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803676
Record Dates: First submitted 2016-01-17; First posted 2016-02-08 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Benign Prostatic Hypertrophy; Lower Urinary Tract Symptoms
Keywords: Prostate Artery Embolization (PAE); Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms (LUTS); PAE; BPH; LUTS; Prostate Artery Embolization; Embospheres
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Embosphere microspheres (Experimental): Embospheres are calibrated microspheres which will be percutaneously delivered intra-arterially via a microcatheter under fluoroscopic guidance to occlude the prostatic arteries.
  Interventions: Device: Embosphere microspheres

INTERVENTIONS:
Device: Embosphere microspheres — This is a clinical trial assessing the feasibly and safety of prostate artery embolization (PAE) for benign prostatic hypertrophy (BPH) resulting in severe lower urinary tract symptoms (LUTS) in patients with gland size ≥90 grams who are TURP ineligible or non-operative candidates with Embosphere microspheres.

SUMMARY:
This is a prospective, open label single center feasibility study to demonstrate basic safety and effectiveness of prostate artery embolization for the treatment of symptomatic benign prostatic Hyperplasia (BPH) in a small series of patients with large (≥90 grams) glands.

DETAILED DESCRIPTION:
This is a prospective, open labeled, non-randomized, single center feasibility study to evaluate the technical and clinical success of prostatic artery embolization utilizing Embosphere microspheres.

At initial consultation patients will be screened to assess the severity of lower urinary tract symptoms (LUTS) related to BPH utilizing the international prostate symptom score (IPSS). After determining eligibility, pre-procedure baseline evaluation will be completed. A baseline prostate ultrasound (TRUS) or MRI will be required to assess prostate mass, and baseline prostate-specific antigen will be measured to help exclude carcinoma and also to follow response to therapy. Patients with suspected malignancy of the prostate will not be enrolled without a negative biopsy finding. Pre- procedure urodynamic studies will be required to assess additional objective measurements and to exclude other causes of LUTS. Cystoscopy will be performed prior to any intervention to help exclude bladder malignancy.

If the patient qualifies by the level of symptoms (IPSS score ≥12), prostate size ≥ 90 grams and max urinary flow rate (Qmax) ≤ 12, the patient will be asked to consider enrolling in the study. A study investigator will review the proposed treatment and baseline/follow-up schedule. If the patient agrees to participate in the study, baseline data will be collected on a case report form and an appointment will be made for prostate artery embolization in the interventional radiology department.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for this study must meet all of the following criteria:

  * Age ≥ 50 years
  * Lower urinary tract symptoms secondary to BPH as defined by:
  * IPSS Symptom Index ≥ 12
  * Maximum Uroflow rate (Qmax) of ≤ 12cc per sec
  * Prostate of ≥ 90 gm as determined by MRI or transrectal ultrasound of the prostate (TRUS)

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from the study.

  * Age less than 50 years
  * Prostate cancer
  * Bladder cancer
  * Severe, life-threatening allergy to iodinated contrast
  * Bilateral internal iliac artery occlusion
  * Causes of obstruction other than BPH such as stricture disease
  * Neurogenic bladder or other causes of bladder atonia
  * Post void residual greater than 250 cc
  * Any contraindication to embolization, including
  * Patients intolerant to occlusion procedures
  * Vascular anatomy or blood flow that precludes catheter placement or embolic agent injection
  * Presence or likely onset of vasospasm
  * Presence or likely onset of hemorrhage
  * Presence of severe atheromatous disease
  * Presence of feeding arteries smaller than distal branches from which they emerge
  * Presence of collateral vessel pathways potentially endangering normal territories during embolization
  * History of any illness or surgery that might confound the results of the study, which produces symptoms that might be confused with those of the disease process under consideration, or which poses additional risk to the patient.
  * Previous prostate surgery, balloon dilatation, stent implantation, laser prostatectomy, hyperthermia, or any other invasive treatment to the prostate
  * Confirmed or suspected bladder cancer
  * Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease
  * Previous pelvic irradiation or radical pelvic surgery
  * Recent (within 3 months) cystolithiasis
  * History or presence of urethral strictures, bladder neck contracture, potentially confounding bladder pathology, or (within 5 years) prostatitis
  * Active urinary tract infection
  * Concomitant medications:

    (i) Use of anti histaminics, anti convulsants, and antispasmodics within 1 week of treatment unless there is documented evidence that the patient has been on the same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study) (ii) Use of alpha blockers, anti-cholinergics, androgens, and gonadotropins-releasing hormonal analogs within 2 months of treatment (iii) Use of 5 alpha reductase inhibitors within 6 months of treatment
  * Compromised renal function (i.e. serum creatinine level greater than 1.8 mg/dl, or upper-tract disease)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12; Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement in Lower Urinary Tract Symptoms (LUTS) | 24 months
  Questionnaire

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 12 months
  Safety and Tolerability as assess by CTCAE 4.0
Change in peak urinary flow (Qmax) | 24 months
  Urodynamics
Change in prostate size | 24 months
  Imaging (MRI or Transrectal ultrasound)
Change in serum PSA from baseline | 24 months
  Blood test
Erectile and sexual function questionnaire | 24 months
  Questionnaire
Pain | 12 months
  Pain Questionnaire
Post void residual bladder volume (PVR) | 24 months
  Imaging (ultrasound)

OTHER OUTCOMES:
Procedural time in minutes | 1 day
  Total PAE time for informational purposes
Total fluoroscopy time in minutes | 1 day
  Total procedural fluoroscopy time in minutes for informational purposes
Size of catheter used for embolization | 1 day
  Microcatheter size for informational purposes
Volume of contrast used in mL | 1 day
  For informational purposes
Length of hospital stay | 1 day
  Expected to be less than 1 day
Volume of embolic material used in mL | 1 day
  Total volume per prostatic artery utilized to achieve stasis
Total fluoroscopy dose mGy | 1 day
  Measured in mGy for informational purposes

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided